CLINICAL TRIAL: NCT01512901
Title: A Randomized, Sham Controlled, Multicenter, Double-Masked, Phase 2/3 Study Assessing Efficacy and Safety of Betamethasone Microsphere in Patients With Macular Edema Following Branch Retinal Vein Occlusion
Brief Title: Efficacy and Safety of Betamethasone Microsphere in Patients With Macular Edema Following Branch Retinal Vein Occlusion (HIKARI)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Santen Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 01021104
Record Dates: First submitted 2012-01-15; First posted 2012-01-19 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Macular Edema Following Branch Retinal Vein Occlusion
MeSH Terms: interventions — salicylhydroxamic acid

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Betamethasone Microsphere (DE-102） Low Dose
- 2 (Experimental)
  Interventions: Drug: Betamethasone Microsphere (DE-102） High Dose
- 3 (Sham Comparator)
  Interventions: Drug: Sham

INTERVENTIONS:
Drug: Betamethasone Microsphere (DE-102） Low Dose
  Arms: 1
Drug: Betamethasone Microsphere (DE-102） High Dose
  Arms: 2
Drug: Sham
  Arms: 3

SUMMARY:
This study will evaluate the efficacy and safety of Betamethasone Microsphere (DE-102) for macular edema following branch retinal vein occlusion

ELIGIBILITY:
Inclusion Criteria:

* 20 years of age or older
* Diagnosis of macular edema following branch retinal vein occlusion

Exclusion Criteria:

* BCVA ETDRS letter score in non-study eye < 35
* Known steroid-responder

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Change from baseline of Best Corrected Visual Acuity(BCVA) in ETDRS letter score

SECONDARY OUTCOMES:
Change in retinal thickness from baseline

CONTACTS AND LOCATIONS:
Locations (2):
- Santen study sites, Osaka, Japan
- Santen study sites, Seoul, South Korea